CLINICAL TRIAL: NCT00111839
Title: Randomized, Phase II, Open-Label Controlled Study of Two Different Doses and Schedules of EMD 72000 (Matuzumab) in Combination With Pemetrexed, or Pemetrexed Alone, as Second-Line Treatment for Stage IIIB/IV Non-Small Cell Lung Cancer and Progressive Disease on or After First-Line Treatment With a Platinum in Combination With Taxanes, Gemcitabine and Vinorelbine
Brief Title: Effects of Matuzumab in Combination With Pemetrexed for the Treatment of Advanced Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD 72000-031; 2006-000899-32 (EudraCT Number)
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer; Non Small Cell Lung Carcinoma
Keywords: Lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; matuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pemetrexed Alone (Active Comparator): Participants will receive pemetrexed 50 milligrams per square meter (mg/m^2) intravenous (IV) infusion every 3 weeks until disease progression (PD) or the occurrence of unacceptable toxicity.
  Interventions: Drug: Pemetrexed
- Pemetrexed Plus Matuzumab 800 mg per Week (Experimental): Participants will receive pemetrexed 50 mg/m^2 IV infusion every 3 weeks in combination with matuzumab 800 milligrams (mg) IV infusion once every week. Treatment will continue until PD or the occurrence of unacceptable toxicity.
  Interventions: Drug: Pemetrexed; Drug: Matuzumab
- Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks (Experimental): Participants will receive pemetrexed 50 mg/m^2 IV infusion every 3 weeks in combination with matuzumab 1600 mg IV infusion every 3 weeks. Treatment will continue until PD or the occurrence of unacceptable toxicity.
  Interventions: Drug: Pemetrexed; Drug: Matuzumab

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed will be administered IV until PD or the occurrence of unacceptable toxicity.
Drug: Matuzumab — Matuzumab will be administered IV until PD or the occurrence of unacceptable toxicity.
  Arms: Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks; Pemetrexed Plus Matuzumab 800 mg per Week

SUMMARY:
This open-label, multicenter, randomized, controlled, Phase II study is planned to answer questions about how the drug, matuzumab (EMD 72000), works and is part of an effort aimed to develop better treatment for advanced lung cancer by combining matuzumab, a monoclonal antibody, with a chemotherapy treatment, called pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided prior to any screening procedure
* Male or female, greater than (>) 18 years of age
* Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC)
* Demonstrated PD on or after first-line chemotherapy for Stage IIIB/IV disease. The first-line therapy must consist of platinum-based regimens in combination with taxanes, gemcitabine or vinorelbine. Stage IIIB/IV participants must have measurable disease (tumor) without clinically significant pleural effusion unless the pleural effusion can be effectively drained prior to admission into the study
* A chemotherapy-free interval of at least 3 weeks between the end of first-line chemotherapy and start of study treatment
* At least 1 measurable lesion according to the modified World Health Organization (WHO) criteria
* Archived tissue or cytologic sample available for the determination of epidermal growth factor receptor (EGFR) expression
* Eastern cooperative oncology group (ECOG) performance status 0-1
* Life expectancy >12 weeks
* Adequate baseline organ functions, defined as: Serum creatinine less than or equal to (≤)1.5*upper limit of normal (ULN). In case of borderline values for serum creatinine, creatinine clearance must be greater than or equal to (≥) 45 millimeters per minute (mL/min); Total bilirubin <1.5*ULN; Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5*ULN (participants with liver metastases should have ALT/AST <5*ULN.); Absolute neutrophil count ≥1500per cubic millimeter(mm^3); Platelet count ≥100000/mm^3; Hemoglobin level ≥10 grams per deciliter
* If procreative potential (male or female), willingness to use effective contraceptive methods for the duration of treatment and continuing for 2 months after the last dose. Participants of procreative potential are defined as any fertile male, or any female who has experienced menarche and who is not postmenopausal (defined as age-related amenorrhea ≥12 months) or who has not undergone successful surgical sterilization (hysterectomy or bilateral oophorectomy)

Exclusion Criteria:

* Radiotherapy or major surgery within 30 days prior to the start of study treatment
* Prior treatment with an EGFR-directed therapy or with EGFR signal transduction inhibitors
* Prior treatment with pemetrexed
* Pregnant (confirmed by beta-human chorionic gonadotropin [β-HCG]) or lactating female
* Weight loss >10% within 12 weeks prior to the start of study treatment
* Documented or symptomatic brain metastases or leptomeningeal disease
* Myocardial infarction within 6 months prior to the start of study treatment, uncontrolled congestive heart failure, or any current New York Heart Association Grade III or IV cardiovascular disorder despite treatment
* Presence of a Grade ≥2 preexisting skin disorder (except for alopecia)
* Previous diagnosis of autoimmune disease with significant organ involvement
* Concurrent malignancies or invasive carcinomas diagnosed within the past 5 years, except for adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix
* Any significant disease that, in the Investigator's opinion, should exclude the participant from the study
* History of significant neurologic or psychiatric disorder (for example, dementia, seizures, or bipolar disorder)
* History of drug abuse within 6 months prior to the start of study treatment
* Known conditions that require concurrent treatment with a nonpermitted drug
* Presence of a contraindication to the study treatment(s) according to the current Investigator's Brochure (IB) for matuzumab and the labeling for pemetrexed
* Known hypersensitivity to the study treatment or any of its components
* Participation in another clinical study within 30 days prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-05-31 (Actual); Primary Completion 2007-07-31 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (58):
- United States (42):
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of Arkansas, Arkansas Cancer Research Center, Little Rock, Arkansas
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Cancer Center or Florida, Ocoee, Florida
  - Peachtree Hematology and Oncology, Atlanta, Georgia
  - Georgia Cancer Specialists, Tucker, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Cancer Institute of Alexian Brothers, Elk Grove Village, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - Hematology-Oncology of Indiana PC, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Kansas City Cancer Center, Overland Park, Kansas
  - Louisville Oncology, Louisville, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - Frederick Memorial Hospital, Frederick, Maryland
  - Tuffs-New England Medical Center, Boston, Massachusetts
  - Henry Ford Health Systems, Detroit, Michigan
  - West Michigan Regional Cancer and Blood Center, Free Soil, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Oncology, Albany, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Presbyterian Hospital Cancer Center, Charlotte, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Dayton Oncology and Hematology, Kettering, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Hematology & Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Mary Crowley Research Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Rainer Oncology Professional Services, Puyallup, Washington
  - Cancer Care Northwest, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
- Austria (4):
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Germany (12):
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Göttingen
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Recklinghausen

REFERENCES:
- [Result] Schiller JH, von Pawel J, Schutt P, Ansari RH, Thomas M, Saleh M, McCroskey RD, Pfeifer W, Marsland TA, Kloecker GH, Sebastian M, Pirker R, Kurek R, Beadman C, Socinski MA. Pemetrexed with or without matuzumab as second-line treatment for patients with stage IIIB/IV non-small cell lung cancer. J Thorac Oncol. 2010 Dec;5(12):1977-85. doi: 10.1097/JTO.0b013e3181f4a5c9. PMID 20978446
- See also: EudraCT results summary synopsis — https://www.clinicaltrialsregister.eu/ctr-search/trial/2006-000899-32/results

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed Alone: Participants received pemetrexed 50 milligrams per square meter (mg/m^2) intravenous (IV) infusion every 3 weeks until disease progression (PD) or the occurrence of unacceptable toxicity.
- Pemetrexed Plus Matuzumab 800 mg Per Week: Participants received pemetrexed 50 mg/m^2 IV infusion every 3 weeks in combination with matuzumab 800 mg IV infusion once every week. An observation period of at least 1 hour was specified between the end of the matuzumab infusion and the start of pemetrexed administration when these treatments were given on the same day. Treatment was continued until PD or the occurrence of unacceptable toxicity.
- Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks: Participants received pemetrexed 50 mg/m^2 IV infusion every 3 weeks in combination with matuzumab 1600 mg IV infusion every 3 weeks. An observation period of at least 1 hour was specified between the end of the matuzumab infusion and the start of pemetrexed administration when these treatments were given on the same day. Treatment was continued until PD or the occurrence of unacceptable toxicity.
Period: Overall Study
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Started | 50 | 51 | 49
Treated | 50 | 51 | 47
Completed | 2 | 5 | 0
Not Completed | 48 | 46 | 49
Not completed — Disease Progression | 30 | 33 | 33
Not completed — Adverse Event | 5 | 3 | 1
Not completed — Protocol Violation | 2 | 4 | 2
Not completed — Death | 1 | 1 | 6
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Logistical Constraint | 1 | 0 | 0
Not completed — Other | 6 | 3 | 3
Not completed — Randomized but Not Treated | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants who received at least one infusion of study treatment.
Groups:
- Pemetrexed Alone: Participants received pemetrexed 50 mg/m^2 IV infusion every 3 weeks until PD or the occurrence of unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks | Total
Number analyzed (Participants) | 50 | 51 | 47 | 148
Age, Continuous [Median (Full Range); unit: years] | 61 [37 to 83] | 62 [48 to 81] | 63 [46 to 78] | 62 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 20 | 53
  Male | 33 | 35 | 27 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Assessed by Independent Review Committee
Description: Objective response was defined as having a complete response (CR) or a partial response (PR). Response assessment was performed using modified World Health Organization (WHO) criteria. Complete response: disappearance of all index and non-index lesions, without appearance of any new lesion. PR: greater than (>) 50 percent (%) decrease from baseline in sum of product of diameters of index lesions, without appearance of any new lesion.
Time Frame: Baseline up to PD or death due to any cause (up to approximately 2 years)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Number analyzed (Participants) | 50 | 51 | 47
participants | 2 [1 to 14] | 8 [7 to 29] | 1 [0 to 11]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from randomization to death (due to any cause). OS was estimated using Kaplan-Meier analysis.
Time Frame: Baseline up to PD or death due to any cause (up to approximately 3.5 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Number analyzed (Participants) | 50 | 51 | 47
months | 7.9 [7.2 to 9.9] | 12.4 [8.8 to NA] — The upper limit of 95% confidence interval (CI) could not be estimated due to insufficient number of participants with event (death). | 5.9 [3.6 to 7.2]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documentation of disease progression (PD) or to death due to any cause, whichever occurred first. PD: >25% increase in one or more lesions, or appearance new lesions. PFS was estimated using Kaplan-Meier analysis.
Time Frame: Baseline up to PD or death due to any cause (up to approximately 3.5 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Number analyzed (Participants) | 50 | 51 | 47
months | 2.7 [1.6 to 4.4] | 2.3 [1.5 to 3.8] | 2.5 [1.4 to 2.9]

4. Secondary Outcome: Duration of Objective Response Assessed by Independent Review Committee
Description: Objective response was defined as having a CR or a PR. Response assessment was performed using modified WHO criteria. CR: disappearance of all index and non-index lesions, without appearance of any new lesion. PR: >50% decrease from baseline in sum of product of diameters of index lesions, without appearance of any new lesion. Duration of objective response was defined as time from first appearance of CR or PR to time of PD (>25% increase in one or more lesions, or appearance new lesions) or death. Duration of objective response was to be assessed using Kaplan-Meier analysis.
Time Frame: From first documented objective response to PD or death due to any cause (up to approximately 3.5 years)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Number analyzed (Participants) | 50 | 51 | 47
months | NA [NA to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | NA [NA to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | NA [NA to NA] — Data could not be estimated due to higher number (>50%) of censored participants.

5. Secondary Outcome: Change From Baseline to Cycle 2 in Global Quality of Life (QoL), as Assessed Using Lung Cancer Symptom Scale (LCSS)
Description: The LCSS consisted of 9 items: 6 items focused on lung cancer symptoms (loss of appetite, fatigue, cough, dyspnea, hemoptysis, and pain] and 3 items were global items (symptom distress, interference with activity level, and global QoL). The global QoL item scores are reported here. The total global QoL item score ranged from 0 (worse QoL) to 100 (best QoL).
Time Frame: Baseline, Cycle 2 (Cycle length = 3 weeks)
Population: ITT population. Here, overall number of participants analyzed = participants with available data for this outcome; number analyzed = participants with available data at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Number analyzed (Participants) | 45 | 46 | 44
units on a scale
  Baseline | 35.9 (26.0) | 31.1 (25.8) | 35.8 (27.5)
  Change at Cycle 2: number analyzed (Participants) | 26 | 25 | 24
  Change at Cycle 2 | 3.5 (17.2) | 0.8 (19.9) | 15.7 (30.7)

ADVERSE EVENTS:
Description: Among SAEs, data for total # affected by any SAE and total # affected by febrile neutropenia are only available. Due diligence was done and all potential information sources have been exhausted; no further information could be retrieved. Hence, for other participants preferred term "Not Available" and System Organ Class "General Disorders" is used.
Arm/Group | Pemetrexed Alone | Pemetrexed Plus Matuzumab 800 mg Per Week | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks
Serious Adverse Events (participants affected / at risk) | 9/50 | 5/51 | 11/47
Other Adverse Events (participants affected / at risk) | 8/50 | 20/51 | 18/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed Alone (N=50) | Pemetrexed Plus Matuzumab 800 mg Per Week (N=51) | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks (N=47)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3
(General disorders) | 8 | 4 | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed Alone (N=50) | Pemetrexed Plus Matuzumab 800 mg Per Week (N=51) | Pemetrexed Plus Matuzumab 1600 mg Every 3 Weeks (N=47)
Neutropenia (Blood and lymphatic system disorders) | 6 | 11 | 7
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Fatigue (General disorders) | 1 | 4 | 1

LIMITATIONS AND CAVEATS:
For serious adverse events (SAEs), due diligence was done and all potential information sources have been exhausted, no further information could be retrieved apart from what is currently reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No